CLINICAL TRIAL: NCT06584253
Title: Relationship of Multidimensional Factors with Digital Addiction Among University Students: a Cross-Sectional Study
Brief Title: Digital Addiction Among University Students
Status: Recruiting | Type: Observational
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, BÜŞRA CANDİRİ, PhD, physiotherapist, Principal Investigator, Inonu University
Other Study IDs: 2024/5922
Record Dates: First submitted 2024-09-02; First posted 2024-09-04 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Internet Addiction; University Student
MeSH Terms: conditions — Internet Addiction Disorder

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Musculoskeletal System Health Questionnaire Scale — It is a 14-item scale that evaluates pain intensity, physical function, sleep, fatigue, emotional state, physical activity level, impact on work and social life, independence, self-management ability and general impact.
Other: International Physical Activity Questionnaire (short form) — International Physical Activity Questionnaire (short form) -
  The IPAQ assesses a range of physical activities, including leisure-time physical activities, indoor and outdoor activities, work-related physical activities, and transportation-related physical activities.
Other: Pittsburgh Sleep Quality Index — It is a questionnaire that evaluates sleep quality with questions asked under 7 main headings: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disorders, use of sleep aids and daytime functions.
Other: Cognitive Failures Questionnaire — The questionnaire aims to measure daily cognitive errors. It assesses simple errors made over the last 6 weeks, as well as perception (e.g., are there times when you can't see something you need at the supermarket even though it's there?), memory (e.g., have you ever forgotten people's names?) and motor functioning (e.g., have you ever bumped into anyone?).
Other: Jamar hand dynamometer — Jamar hand dynamometer - students will perform grip strength assessments with their dominant hand while seated. As recommended by the American Association of Hand Therapists protocol, students will sit in a comfortable chair with their shoulders neutrally rotated and adducted, elbow flexed to 90°, and wrist and forearm in neutral positions.
Other: Depression Anxiety Stress Scale - 21 Short Form — DASÖ-21 consists of 3 subcategories (depression, anxiety and stress). Each category consists of 7 separate questions and a total of 21 questions.
Other: Body Awareness Questionnaire — The questionnaire aims to determine the level of body composition sensitivity.
Other: SF-12 — This questionnaire consists of two general components related to physical and mental function, consisting of 12 questions and 8 scales measuring physical function (2 questions), bodily pain (1 question), role limitations due to physical problems (2 questions), general health (1 question) vitality (40).

SUMMARY:
The aim of this study is to contribute to our understanding of digital media addiction by investigating the prevalence of digital addiction among university students and examining the relationship between variables such as body awareness, physical activity levels, hand grip strength, upper extremity function and pain-dash, quality of life, depression, stress, anxiety, sleep quality, and cognitive levels and digital addiction.

DETAILED DESCRIPTION:
After recording the demographic information of all individuals participating in the study, screen addiction, BMI, body awareness, physical activity levels, handgrip strength, upper extremity pain and function and pain-dash, quality of life, depression, stress, anxiety, sleep quality, cognitive levels will be evaluated. Individuals will be asked to fill out self-report questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* University students aged 18 and over
* Those who have been using smartphones for more than a year

Exclusion Criteria:

* People under the age of 18,
* Those diagnosed by a doctor with any musculoskeletal, rheumatic, neurological, cardiovascular system diseases or diagnosed with a mental disorder, sleep disorder such as narcolepsy or addiction to alcohol, substances, etc.
* Those with any history of injury or surgery in the upper extremity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: University students
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2024-05-21 (Actual); Primary Completion 2024-09-12 (Estimated); Study Completion 2024-09-12 (Estimated)

PRIMARY OUTCOMES:
Musculoskeletal System Health Questionnaire Scale | 24-48 hours
  It is a 14-item scale that evaluates pain intensity, physical function, sleep, fatigue, emotional state, physical activity level, impact on work and social life, independence, self-management ability and general impact.Each Question is scored from 0-4. Higher scores indicate better MSK health status.
International Physical Activity Questionnaire (short form) | 24-48 hours
  The IPAQ assesses a range of physical activities, including leisure-time physical activities, indoor and outdoor activities, work-related physical activities, and transportation-related physical activities.
Pittsburgh Sleep Quality Index | 24-48 hours
  It is a questionnaire that evaluates sleep quality with questions asked under 7 main headings: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disorders, use of sleep aids and daytime functions.Higher overall scores indicate poorer sleep quality
Cognitive Failures Questionnaire | 24-48 hours
  The questionnaire aims to measure daily cognitive errors. It assesses simple errors made over the last 6 weeks, as well as perception (e.g., are there times when you can't see something you need at the supermarket even though it's there?), memory (e.g., have you ever forgotten people's names?) and motor functioning (e.g., have you ever bumped into anyone?).The total score ranges from 0 to 100. High scores indicate an increased tendency for cognitive failure.
Jamar hand dynamometer | 24-48 hours
  Jamar hand dynamometer - students will perform grip strength assessments with their dominant hand while seated. As recommended by the American Association of Hand Therapists protocol, students will sit in a comfortable chair with their shoulders neutrally rotated and adducted, elbow flexed to 90°, and wrist and forearm in neutral positions.
Depression Anxiety Stress Scale - 21 Short Form | 24-48 hours
  DASÖ-21 consists of 3 subcategories (depression, anxiety and stress). Each category consists of 7 separate questions and a total of 21 questions.Higher scores indicate more severe emotional distress
Body Awareness Questionnaire | 24-48 hours
  The questionnaire aims to determine the level of body composition sensitivity.The survey consists of 18 statements and participants are asked to rate each statement on a scale of 1-7. A higher score indicates better body awareness.
SF-12 | 24-48 hours
  This questionnaire consists of two general components related to physical and mental function, consisting of 12 questions and 8 scales measuring physical function (2 questions), bodily pain (1 question), role limitations due to physical problems (2 questions), general health (1 question) vitality (40).Scoring ranges from 0 to 100, with higher scores indicating better quality of life.
Digital Addiction Scale | 24-48 hours
  The Digital Addiction Scale (DAS) was used to assess the participants' digital addiction levels. The scale consists of 19 questions with 5 sub-factors (excessive use, deprivation, disruption of life flow, emotional state and addiction). The total score is between 19-95, with a high score indicating a high level of media addiction.

CONTACTS AND LOCATIONS:
Overall Officials: dilan demirtas karaoba, asst. prof, Study Director — Inonu University
Locations (2):
- Turkey (Türkiye) (2):
  - Dilan Demirtas Karaoba, Iğdır, Iğdır
  - Dilan, Iğdır, Iğdır

IPD SHARING:
Plan to Share IPD: No